CLINICAL TRIAL: NCT02566070
Title: COntinuous vs BOlus Nasogastric Feeding in Mechanically Ventilated Pediatric Patients 2
Acronym: COBO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150311
Record Dates: First submitted 2015-09-24; First posted 2015-10-01 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Dietary Modification
Keywords: Enteral feeding; Continuous gastric feeding; Bolus gastric feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Gastric Feeding (CGF) (Active Comparator): CGF group will have total daily enteral nutrition requirement delivered at a constant rate via infusion over the entire 24 hour period.
  Interventions: Other: Continuous Gastric Feeding
- Bolus Gastric Feeding (BGF) (Experimental): BGF group will have total daily enteral nutrition requirement delivered in interval, finite volumes over the course of the 24 hour period.
  Interventions: Other: Bolus Gastric Feeding

INTERVENTIONS:
Other: Continuous Gastric Feeding
  Arms: Continuous Gastric Feeding (CGF)
Other: Bolus Gastric Feeding
  Arms: Bolus Gastric Feeding (BGF)

SUMMARY:
This multi-center, prospective, randomized comparative effectiveness intervention study will evaluate continuous feeding (CGF) and bolus gastric feeding (BGF) protocols and their effect on delivery of prescribed nutrition and feeding intolerance in mechanically ventilated critically ill children for up through 12 hours post achievement goal feeds or exclusion from feeding protocol, whichever comes first, to a maximum of 10 days.

DETAILED DESCRIPTION:
A significant number of children (>30%) are malnourished upon admission to the Pediatric Intensive Care Unit (PICU). In addition, critically ill children are at risk to develop new or worsened malnutrition during their PICU stay. Adequate nutritional support of critically ill children reduces mortality and morbidities, such as hospital acquired health care infections. Inadequate nutrition during hospitalization results in poor healing, increased risk for hospital acquired conditions, and prolonged length of stay, all of which contribute to increased health care costs. Even previously healthy children experiencing critical illness are at high risk for malnourishment because of increased protein and/or caloric needs at a time when oral intake is inadequate to meet their metabolic needs. A gap in the literature exists regarding the effectiveness of 2 delivery modes for gastric enteral nutrition: continuous gastric (stomach) feeding (CGF), the steady infusion of liquid nutrition is delivered at an hourly volume via an infusion pump, and bolus gastric feeding (BGF), whereby nutrition is intermittently delivered over a prescribed period of time, followed by a period of rest.

Enteral nutrition (EN, or tube feeding) in the PICU is commonly given via continuous gastric feeding. However, feeding by bolus or intermittent methods better mimics normal body function and may minimize interruptions to feedings improving nutritional intake. This study proposes to address the gap in the literature regarding the best method to deliver EN to achieve prescribed nutritional goals and avoid feeding interruptions in the mechanically ventilated, critically ill pediatric population.

This multi-center, prospective, randomized, controlled study includes children 1-month to 12-years who are on a ventilator and have EN started within 48-hours of admission. Subjects are randomized to CGF or BGF. Feeding volume is advanced in a weight-based manner every 3-hours to target volume; caloric density is then increased to goal. Feeding intolerance measures are assessed every 3-hours. Study sites are assigned to follow one of two feeding intolerance criteria to better define the measures and thresholds necessary to halt and resume feeds for safety purposes. Incidence, duration and category of feeding interruptions are recorded. Statistical significance is defined as p < 0.05. The findings will be submitted for oral and poster presentation and manuscripts submitted for publication.

As the focus of nursing remains not on disease and cure, rather on healing and health, nutrition is embedded in this philosophy. Our vision of nursing is to put the patient in the best position to heal him or herself. Mitigating existing malnutrition and/or avoiding newly acquired nutritional deficits decreases the risk of mortality and hospital acquired adverse events in this population. This study seeks to optimize delivery of nutrition as therapy as imperative to optimize clinical and functional outcomes in the critically ill child.

ELIGIBILITY:
Inclusion Criteria:

* all medical patients hospitalized in the Pediatric Intensive Care Unit (PICU)
* aged 1 month through 12 years of age
* mechanically ventilated within the first 24 hours of admission
* patients with an anticipated duration of mechanical ventilation greater than 48 hours

Exclusion Criteria:

* diagnosis of acute or chronic gastrointestinal pathology
* primary cardiac surgery or other surgical service patients
* enteral nutrition initiated greater than 48 hours post PICU admission, or
* enteral nutrition was initiated prior to admission to PICU

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Time to goal feeds (TTGF) is decreased in a bolus compared to continuous gastric feeding protocol. | 12 to 48 hours post enteral feeding
  TTGF defined as time to attain goal feeds

SECONDARY OUTCOMES:
Feeding interruptions | 12 to 48 hours post enteral feeding
  measured by minutes feeds are withheld.
Gastric residual volumes | 12 to 48 hours post enteral feeding
  measured in milliliters
Rate of ventilator associated infections (VAI) | 12 to 48 hours post enteral feeding
  as reported by Infection Control Department.
Oxygen Saturation Index | 12 to 48 hours post enteral feeding
  as calculated by [(FiO2 x Mean Airway Pressure)/SpO2]
Emesis | 12 to 48 hours post enteral feeding
  as a binary yes/no event
Abdominal girth | 12 to 48 hours post enteral feeding
  measured in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie Brown, PhD, CPNP, Principal Investigator — Akron Children's Hospital
Locations (6):
- United States (6):
  - Shands Children's Hospital, Gainesville, Florida
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - The Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta NM, Bechard LJ, Cahill N, Wang M, Day A, Duggan CP, Heyland DK. Nutritional practices and their relationship to clinical outcomes in critically ill children--an international multicenter cohort study*. Crit Care Med. 2012 Jul;40(7):2204-11. doi: 10.1097/CCM.0b013e31824e18a8. PMID 22564954
- [Background] Mikhailov TA, Kuhn EM, Manzi J, Christensen M, Collins M, Brown AM, Dechert R, Scanlon MC, Wakeham MK, Goday PS. Early enteral nutrition is associated with lower mortality in critically ill children. JPEN J Parenter Enteral Nutr. 2014 May;38(4):459-66. doi: 10.1177/0148607113517903. Epub 2014 Jan 8. PMID 24403379
- [Background] Mehta NM, McAleer D, Hamilton S, Naples E, Leavitt K, Mitchell P, Duggan C. Challenges to optimal enteral nutrition in a multidisciplinary pediatric intensive care unit. JPEN J Parenter Enteral Nutr. 2010 Jan-Feb;34(1):38-45. doi: 10.1177/0148607109348065. Epub 2009 Nov 10. PMID 19903872
- [Background] Khorasani EN, Mansouri F. Effect of early enteral nutrition on morbidity and mortality in children with burns. Burns. 2010 Nov;36(7):1067-71. doi: 10.1016/j.burns.2009.12.005. Epub 2010 Apr 18. PMID 20403667
- [Background] Schindler CA, Mikhailov TA, Kuhn EM, Christopher J, Conway P, Ridling D, Scott AM, Simpson VS. Protecting fragile skin: nursing interventions to decrease development of pressure ulcers in pediatric intensive care. Am J Crit Care. 2011 Jan;20(1):26-34; quiz 35. doi: 10.4037/ajcc2011754. PMID 21196569
- [Background] Larsen BM, Goonewardene LA, Field CJ, Joffe AR, Van Aerde JE, Olstad DL, Clandinin MT. Low energy intakes are associated with adverse outcomes in infants after open heart surgery. JPEN J Parenter Enteral Nutr. 2013 Mar;37(2):254-60. doi: 10.1177/0148607112463075. Epub 2012 Oct 11. PMID 23064254
- [Background] Mehta NM, Compher C; A.S.P.E.N. Board of Directors. A.S.P.E.N. Clinical Guidelines: nutrition support of the critically ill child. JPEN J Parenter Enteral Nutr. 2009 May-Jun;33(3):260-76. doi: 10.1177/0148607109333114. No abstract available. PMID 19398612
- [Background] Brown A-M, Forbes ML, Vitale VS, Tirodker UH, Zeller R. Effects of a gastric feeding protocol on efficiency of enteral nutrition in critically ill infants and children. ICAN: Infant, Child, & Adolescent Nutrition. 2012;4(3):175-180.
- [Background] Tume L, Carter B, Latten L. A UK and Irish survey of enteral nutrition practices in paediatric intensive care units. Br J Nutr. 2013 Apr 14;109(7):1304-22. doi: 10.1017/S0007114512003042. Epub 2012 Aug 1. PMID 22853808
- [Background] Mohr F, Steffen R. Physiology of gastrointestinal motility. In: Wyllie R, Hyams JS, Kay M, eds. Pediatric Gastrointestinal and Liver Disease. 4th ed. Philadelphia, PA: Elsevier/Saunders; 2011:39-49.
- [Background] Chen YC, Chou SS, Lin LH, Wu LF. The effect of intermittent nasogastric feeding on preventing aspiration pneumonia in ventilated critically ill patients. J Nurs Res. 2006 Sep;14(3):167-80. doi: 10.1097/01.jnr.0000387575.66598.2a. PMID 16967399
- [Background] Lee JS, Auyeung TW. A comparison of two feeding methods in the alleviation of diarrhoea in older tube-fed patients: a randomised controlled trial. Age Ageing. 2003 Jul;32(4):388-93. doi: 10.1093/ageing/32.4.388. PMID 12851181
- [Background] Lee JS, Kwok T, Chui PY, Ko FW, Lo WK, Kam WC, Mok HL, Lo R, Woo J. Can continuous pump feeding reduce the incidence of pneumonia in nasogastric tube-fed patients? A randomized controlled trial. Clin Nutr. 2010 Aug;29(4):453-8. doi: 10.1016/j.clnu.2009.10.003. Epub 2009 Nov 12. PMID 19910085
- [Background] Horn D, Chaboyer W. Gastric feeding in critically ill children: a randomized controlled trial. Am J Crit Care. 2003 Sep;12(5):461-8. PMID 14503430
- [Background] Hurt RT, McClave SA. Gastric residual volumes in critical illness: what do they really mean? Crit Care Clin. 2010 Jul;26(3):481-90, viii-ix. doi: 10.1016/j.ccc.2010.04.010. PMID 20643301
- [Background] Skillman HE. Monitoring the efficacy of a PICU nutrition therapy protocol. JPEN J Parenter Enteral Nutr. 2011 Jul;35(4):445-6. doi: 10.1177/0148607111409046. Epub 2011 Jun 1. No abstract available. PMID 21632953
- [Background] Reignier J, Mercier E, Le Gouge A, Boulain T, Desachy A, Bellec F, Clavel M, Frat JP, Plantefeve G, Quenot JP, Lascarrou JB; Clinical Research in Intensive Care and Sepsis (CRICS) Group. Effect of not monitoring residual gastric volume on risk of ventilator-associated pneumonia in adults receiving mechanical ventilation and early enteral feeding: a randomized controlled trial. JAMA. 2013 Jan 16;309(3):249-56. doi: 10.1001/jama.2012.196377. PMID 23321763
- [Background] Skillman HE. How you can improve the delivery of enteral nutrition in your PICU. JPEN J Parenter Enteral Nutr. 2010 Jan-Feb;34(1):99-100. doi: 10.1177/0148607109344725. No abstract available. PMID 20054060
- [Background] Weckwerth JA. Monitoring enteral nutrition support tolerance in infants and children. Nutr Clin Pract. 2004 Oct;19(5):496-503. doi: 10.1177/0115426504019005496. PMID 16215145
- [Background] Horn D, Chaboyer W, Schluter PJ. Gastric residual volumes in critically ill paediatric patients: a comparison of feeding regimens. Aust Crit Care. 2004 Aug;17(3):98-100, 102-3. doi: 10.1016/s1036-7314(04)80011-0. PMID 15493856
- [Background] Cooper VB, Haut C. Preventing ventilator-associated pneumonia in children: an evidence-based protocol. Crit Care Nurse. 2013 Jun;33(3):21-9; quiz 30. doi: 10.4037/ccn2013204. PMID 23727849
- [Background] Thomas NJ, Shaffer ML, Willson DF, Shih MC, Curley MA. Defining acute lung disease in children with the oxygenation saturation index. Pediatr Crit Care Med. 2010 Jan;11(1):12-7. doi: 10.1097/PCC.0b013e3181b0653d. PMID 19561556
- [Background] Poulard F, Dimet J, Martin-Lefevre L, Bontemps F, Fiancette M, Clementi E, Lebert C, Renard B, Reignier J. Impact of not measuring residual gastric volume in mechanically ventilated patients receiving early enteral feeding: a prospective before-after study. JPEN J Parenter Enteral Nutr. 2010 Mar-Apr;34(2):125-30. doi: 10.1177/0148607109344745. Epub 2009 Oct 27. PMID 19861528
- [Background] Ukleja A. Altered GI motility in critically Ill patients: current understanding of pathophysiology, clinical impact, and diagnostic approach. Nutr Clin Pract. 2010 Feb;25(1):16-25. doi: 10.1177/0884533609357568. PMID 20130154
- [Background] Brown A-M. A Comparison of Two Gastric Feeding Approaches in Mechanically Ventilated Pediatric Patients. Akron, OH: The University of Akron; 2014:159.